CLINICAL TRIAL: NCT03300505
Title: ARRO-CITO: (UMCC 2017.055) Phase Ib/II Single-Arm Multi-Center Study of IONIS-AR-2.5Rx, a Next Generation Androgen Receptor Antisense Oligonucleotide, in Combination With Enzalutamide in Metastatic Castration Resistant Prostate Cancer
Brief Title: ARRx in Combination With Enzalutamide in Metastatic Castration Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Cancelled by the sponsor
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2017.055; HUM00130051 (Other: University of Michigan); 5P50CA186786-10 (NIH)
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARRx + Enzalutamide (Experimental): Phase 1b: All registered subjects will be treated with ARRx (ASO) in combination with enzalutamide. ARRx will be given intravenously on Days 1, 4, 8, 11, 15 on cycle 1, then on days 1, 8, 15 in subsequent 21-day cycles. Enzalutamide will be taken daily in 21 day cycles starting Day 1 of cycle 1. Treatment will continue until clinical or radiologic progression or unacceptable toxicity.
  Phase 2: Subjects will be treated with ARRx (ASO) at the maximum tolerated (MTD), in combination with enzalutamide until clinical or radiologic progression or unacceptable toxicity. (Schedule of administration as in phase 1b.)
  Interventions: Drug: ARRx; Drug: Enzalutamide

INTERVENTIONS:
Drug: ARRx — Given intravenously (IV)
  Other Names: AZD5312
Drug: Enzalutamide — Given by mouth (PO)
  Other Names: Xtandi

SUMMARY:
The purpose of this study is to test the effectiveness (how well the drug works), safety, and tolerability of the investigational drug combination of ARRx (also known as AZD5312) plus enzalutamide in patients with metastatic castration resistant prostate cancer.

DETAILED DESCRIPTION:
This is a single dose-finding one-arm phase Ib/II trial to determine the maximum tolerated dose (MTD) from among three dose levels of ARRx in combination with a fixed dose of enzalutamide and to obtain a preliminary estimate of efficacy at this MTD, as measured by PSA response rate. Success for the trial is defined as finding a dose level that is likely to be both tolerable and effective.

The study was originally registered as a phase 1/ phase 2 study; however, the study was cancelled by the sponsor before opening the phase 2 portion. Outcome measures were updated to include those relevant to the Phase 1 portion as the study was terminated before enrolling into phase 2

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and voluntarily agree to participate by providing written informed consent for the trial.
* Histologically confirmed prostate adenocarcinoma cancer, either pure or mixed. Small cell/neuroendocrine differentiation is not allowed.
* Castrate levels of serum testosterone (≤ 50 ng/dL). Patients must continue androgen deprivation therapy with an LHRH analogue or antagonist if they have not undergone bilateral orchiectomy.
* Patients must have metastatic disease; either non-measurable disease OR measurable disease per RECIST 1.1.
* Progressive disease despite ongoing treatment with Androgen Deprivation Therapy (ADT).
* Patients treated with first generation anti-androgen as most recent systemic therapy (e.g. bicalutamide, nilutamide) must have at least 4 weeks elapsed from treatment discontinuation to start of protocol therapy with evidence of disease progression (per protocol) following discontinuation of prior anti-androgen.
* Minimum PSA at entry of 1 ng/mL is required.
* ECOG Performance Status 0, 1 or 2.
* Be ≥18 years of age on the day of signing informed consent.
* Demonstrate adequate organ function.
* Subjects must agree to use an adequate method of contraception as outlined in the protocol starting with the time of informed consent through 120 days after the last dose trial therapy.

Exclusion Criteria:

* Prior chemotherapy and/or enzalutamide for metastatic castration-resistant prostate cancer. Chemotherapy administered in the castration-sensitive setting is allowed provided last dose of chemotherapy was greater than 6 months prior to study entry.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigation device within 4 weeks prior to enrollment.
* Has not recovered (i.e., AE ≤Grade 1 or at baseline) from AEs due to a previously administered agent. Subjects with ≤Grade 2 neuropathy or ≤Grade 2 alopecia are an exception to this criterion and are allowed if relevant toxicity is stabilized.
* If subjects received major surgery they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting trial therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial. At the time of signing informed consent is a known regular user (including "recreational use") of any illicit drug(s) or had a recent history (within the last year) of drug or alcohol abuse.
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
* Has known active hepatitis B (e.g., HBsAg reactive) or hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live virus vaccine within 30 days of planned start of trial therapy.
* Has known active CNS metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they have stable brain metastases (stability is normally defined as a period of 1 to 3 months in which there is no evidence of new or enlarging CNS metastases).
* Has symptomatic ascites or pleural effusion; a subject who is clinically stable following treatment for these conditions is eligible.
* Has had a prior allogeneic stem cell or bone marrow transplant.
* Has known contraindication to aspirin (81 mg).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajjai Alva, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: 600 mg IONIS; Dose Level 2: 750 mg IONIS; Dose Level 3: 900 mg IONIS: Phase 1b: All registered subjects will be treated with ARRx (ASO) in combination with enzalutamide. ARRx will be given intravenously on Days 1, 4, 8, 11, 15 on cycle 1, then on days 1, 8, 15 in subsequent 21-day cycles. Enzalutamide will be taken daily in 21 day cycles starting Day 1 of cycle 1. Treatment will continue until clinical or radiologic progression or unacceptable toxicity.
  ARRx: Given intravenously (IV)
  Enzalutamide: Given by mouth (PO)
  Dose Level 1: 600 mg IONIS Dose Level 2: 750 mg IONIS Dose Level 3: 900 mg IONIS
Period: Overall Study
Arm/Group | Dose Level 1: 600 mg IONIS | Dose Level 2: 750 mg IONIS | Dose Level 3: 900 mg IONIS
Started | 1 | 5 | 3
Completed | 1 | 2 | 0
Not Completed | 0 | 3 | 3
Not completed — Death | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Sponsor Termination | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Only a single participant was included in the Dose Level 1 arm and data are not reported publicly to protect participant confidentiality
Groups:
- Dose Level 1; Dose Level 2; Dose Level 3: Phase 1b: All registered subjects will be treated with ARRx (ASO) in combination with enzalutamide. ARRx will be given intravenously on Days 1, 4, 8, 11, 15 on cycle 1, then on days 1, 8, 15 in subsequent 21-day cycles. Enzalutamide will be taken daily in 21 day cycles starting Day 1 of cycle 1. Treatment will continue until clinical or radiologic progression or unacceptable toxicity.
  ARRx: Given intravenously (IV) Enzalutamide: Given by mouth (PO) Dose Level 1: 600 mg IONIS
  Dose Level 2: 750 mg IONIS
  Dose Level 3: 900 mg IONIS
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Total
Number analyzed (Participants) | 1 | 5 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants] — Population: Only a single participant was included in the Dose Level 1 arm and data are not reported publicly to protect participant confidentiality
  Participants
    number analyzed (Participants) | 0 | 5 | 3 | 8
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 0 | 1 | 1 | 2
    >=65 years | 0 | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only a single participant was included in the Dose Level 1 arm and data are not reported publicly to protect participant confidentiality
  Participants
    number analyzed (Participants) | 0 | 5 | 3 | 8
    Female | 0 | 0 | 0 | 0
    Male | 0 | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only a single participant was included in the Dose Level 1 arm and data are not reported publicly to protect participant confidentiality
  Participants
    number analyzed (Participants) | 0 | 5 | 3 | 8
    Hispanic or Latino | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 0 | 5 | 3 | 8
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only a single participant was included in the Dose Level 1 arm and data are not reported publicly to protect participant confidentiality
  Participants
    number analyzed (Participants) | 0 | 5 | 3 | 8
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 1 | 1 | 2
    White | 0 | 4 | 2 | 6
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: Only a single participant was included in the Dose Level 1 arm and data are not reported publicly to protect participant confidentiality
  participants
    United States: number analyzed (Participants) | 0 | 5 | 3 | 8
    United States |  | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Dose-limiting Toxicity (DLT) During the First Cycle of ARRx (in Combination With Enzalutamide)
Description: DLTs will be counted based on the number of subjects with DLT at a given dose level. No single subject can trigger more than one DLT event. DLT is defined as any Grade 3 or higher toxicity as defined by CTCAE v5.0. Toxicity that is clearly and directly related to the primary disease or to another etiology is excluded from this definition.
Time Frame: Up to day 21 of treatment
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Level 1; Level 2; Level 3: Phase 1b: All registered subjects will be treated with ARRx (ASO) in combination with enzalutamide. ARRx will be given intravenously on Days 1, 4, 8, 11, 15 on cycle 1, then on days 1, 8, 15 in subsequent 21-day cycles. Enzalutamide will be taken daily in 21 day cycles starting Day 1 of cycle 1. Treatment will continue until clinical or radiologic progression or unacceptable toxicity.
  ARRx: Given intravenously (IV) Enzalutamide: Given by mouth (PO) Dose Level 1: 600 mg IONIS Dose Level 2: 750 mg IONIS Dose Level 3: 900 mg IONIS
Arm/Group | Level 1 | Level 2 | Level 3
Number analyzed (Participants) | 0 | 5 | 3
Participants |  | 0 | 0

2. Primary Outcome: Best PSA Response
Description: Number of subjects with at least 50% decline in PSA from Baseline
Time Frame: 3.5 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Level 1 | Level 2 | Level 3
Number analyzed (Participants) | 0 | 5 | 3
Participants |  | 4 | 3

3. Secondary Outcome: Percentage of Patients With a Reduction in PSA of at Least 30% From Baseline
Description: Using PCWG3 criteria. Number of patient with a reduction in PSA of at least 30% from baseline
Time Frame: 3.5 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Level 1 | Level 2 | Level 3
Number analyzed (Participants) | 0 | 5 | 3
Participants |  | 4 | 3

4. Secondary Outcome: Overall Survival at One Year
Description: One year KM estimate. Patients alive or lost to follow-up at the time of analysis will be censored at their last date of follow-up.
Time Frame: 1 year
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Level 1 | Level 2 | Level 3
Number analyzed (Participants) | 0 | 5 | 3
percentage of participants |  | 67 [5 to 95] | 100 [100 to 100]

5. Secondary Outcome: Intrapatient Dose Delays
Description: Number of participants that experienced dose delays while on study treatment
Time Frame: 3.5 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Level 1 | Level 2 | Level 3
Number analyzed (Participants) | 0 | 5 | 3
Participants |  | 3 | 3

6. Secondary Outcome: Intrapatient Dose Reductions
Description: Number of participants that experienced dose reductions while on study treatment
Time Frame: 3.5 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Level 1 | Level 2 | Level 3
Number analyzed (Participants) | 0 | 5 | 3
Participants |  | 1 | 1

ADVERSE EVENTS:
Time Frame: All adverse event data (serious and non-serious) collected from the time of the initial study treatment administration through 30 days after the last dose of study treatment; additionally, any serious adverse event occurring more than 30 days after the last study treatment if considered to be related to the study treatment. Data was collected during a 3.5 year period.
Description: Only a single participant was included in the Dose Level 1 arm and data are not reported publicly to protect participant confidentiality
Arm/Group | Level 1 | Level 2 | Level 3
All-Cause Mortality (participants affected / at risk) | 0/0 | 1/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 2/5 | 1/3
Other Adverse Events (participants affected / at risk) | 0/0 | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Level 1 (N=1) | Level 2 (N=5) | Level 3 (N=3)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic Event (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Sepsis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Level 1 (N=0) | Level 2 (N=5) | Level 3 (N=3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 3 (5)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 3 (4) | 2 (2)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (4) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 3 (5)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT03300505/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT03300505/ICF_001.pdf